CLINICAL TRIAL: NCT05478928
Title: Effects of Invasive Techniques in Myofascial Trigger Points: A Randomized Controlled Clinical Trial
Brief Title: Invasive Techniques in Trigger Points
Acronym: ITTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimonides University (Other)
Responsible Party: Principal Investigator, Oscar Ronzio, Head of Physiotherapy program, Maimonides University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 863
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Trigger point; Percutaneous; Electrolysis; Physical Therapy Modalities
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dynamic dry needling (Experimental): Dynamic dry needling will be done in the upper trapezius trigger point.
  Interventions: Other: Dynamic dry needling
- Fixed dose dynamic MEP (Experimental): Dynamic low intensity percutaneous electrolysis will be applied in the upper trapezius trigger point with a fixed dose.
  Interventions: Device: Fixed dose dynamic MEP
- Static dry needling: (Experimental): Static dry needling will be done in the upper trapezius trigger point.
  Interventions: Other: Static Dry needling
- Fixed dose static MEP (Experimental): Static low intensity percutaneous electrolysis will be applied in the upper trapezius trigger point with a fixed dose.
  Interventions: Device: Fixed dose static MEP
- Algorithm-based dose static MEP (Experimental): Low intensity percutaneous electrolysis will be applied in the upper trapezius trigger point with an algorithm-based dose.
  Interventions: Device: Algorithm-based dose static MEP
- Placebo (Placebo Comparator): An acupuncture needle will be slightly introduced into the upper trapezius trigger point.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Dynamic dry needling — An acupuncture needle of 0.3 x 25 mm will be introduced perpendicularly into the upper trapezius trigger point. A movement with the needle will be done at 1 Hz for 120 seconds.
  Arms: Dynamic dry needling
Device: Fixed dose dynamic MEP — Cathodic low intensity percutaneous electrolysis will be applied through an acupuncture needle of 0.3 x 25 mm in the upper trapezius trigger point. A movement with the needle will be done at 1 Hz with an intensity of 600 micro-Amperes. If the patient refers discomfort, the procedure will be stopped and resumed totalling 120 seconds (total dose of 72 mC).
  Arms: Fixed dose dynamic MEP
Other: Static Dry needling — An acupuncture needle of 0.3 x 25 mm will be introduced perpendicularly into the upper trapezius trigger point for 120 seconds.
  Arms: Static dry needling:
Device: Fixed dose static MEP — Cathodic low intensity percutaneous electrolysis will be applied through an acupuncture needle of 0.3 x 25 mm in the upper trapezius trigger point. The therapy will be done statically with an intensity of 600 micro-Amperes. If the patient refers discomfort, the procedure will be stopped and resumed totalling 120 seconds (total dose of 72 mC).
  Arms: Fixed dose static MEP
Device: Algorithm-based dose static MEP — Cathodic low intensity percutaneous electrolysis will be applied through an acupuncture needle of 0.3 x 25 mm in the upper trapezius trigger point. The therapy will be done statically, at 600 micro-Amperes. If the patient refers discomfort, the procedure will be stopped and resumed. Treatment will finish when the patient does not refer any discomfort for a period longer than 60 seconds. Total dose in mC will be registered.
  Arms: Algorithm-based dose static MEP
Other: Placebo — An acupuncture needle of 0.3 x 25 mm will be introduced perpendicularly up to 3 mm deep into the upper trapezius trigger point for 120 seconds.
  Arms: Placebo

SUMMARY:
Myofascial pain syndrome (MPS) is present in up to 87% of the patients that present pain. MPS usually presents painful myofascial trigger points (MTrPs).

One methodology used to quantify the pain in MPS is the algometry, which measures the pressure pain threshold (PPT).

Invasive techniques in physiotherapy have become popular in the last years due to their clinical efficacy and evidence. Percutaneous Microelectrolysis (MEP®) and dry needling are techniques that are already in use for this syndrome.

MEP® is a technique that employs a galvanic current up to 990 microAmperes, which is applied percutaneously with an acupuncture needle connected to the cathode. It is also known as low intensity percutaneous electrolysis.

The aim of this study is to compare the effects in pain and muscle tone (measured with algometry and surface electromyography) of invasive techniques. Healthy subjects between 18 to 48 years old, both sex, presenting MTrPs in upper trapezius will be recruited.

The secondary objectives are to determine the discomfort degree of each technique and if it is better to use MEP® with a fixed dose or with an algorithm in which the dose varies.

The hypothesis, according to our previous studies, is that MEP® generates higher changes in PPT.

ELIGIBILITY:
Inclusion Criteria:

1. Neck pain during the last 6 months
2. Presence of a palpable taut band in the upper trapezius
3. Presence of a hypersensitive tender spot in the taut band, with local or referred pain elicitation in response to compression
4. PPT less than 3 Kg/cm2

Exclusion Criteria:

1. Previous cervical and/or shoulder surgical intervention.
2. Phobia to needles.
3. Temporomandibular disorders.
4. Medicated with anticoagulants
5. Still receiving a treatment for the myofascial trigger points (Physical therapy, NSAIDs, etc.)
6. Diagnosis of fibromyalgia.
7. Radiculopathies and/or radicular pain
8. Whiplash related neck pain
9. Migraines
10. Dizziness
11. Endocrinal diseases
12. Being pregnant
13. Cancer

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) - Baseline | Baseline
  Algometry is used to measure the Pressure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It will be applied in the Myofascial Trigger points.
Pressure Pain Threshold (PPT) - 10 minutes | 10 minutes
  Algometry is used to measure the Pressure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It will be applied in the Myofascial Trigger points.
Pressure Pain Threshold (PPT) - 24 hours | 24 hours
  Algometry is used to measure the Pressure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It will be applied in the Myofascial Trigger points.
Pressure Pain Threshold (PPT) - 48 hours | 48 hours
  Algometry is used to measure the Pressure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It will be applied in the Myofascial Trigger points.
Pressure Pain Threshold (PPT) - Day 7 | Day 7
  Algometry is used to measure the Pressure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It will be applied in the Myofascial Trigger points.
Surface electromyography at rest - Baseline | Baseline
  Electromyography (EMG) is used to measure muscular electrical activity at rest to determine the basal tone. Peak voltage and root mean square (RMS) voltage will be informed.
Surface electromyography at rest - 10 minutes | 10 minutes
  Electromyography (EMG) is used to measure muscular electrical activity at rest to determine the basal tone. Peak voltage and root mean square (RMS) voltage will be informed.
Surface electromyography at rest - 24 hours | 24 hours
  Electromyography (EMG) is used to measure muscular electrical activity at rest to determine the basal tone. Peak voltage and root mean square (RMS) voltage will be informed.
Surface electromyography at rest - 48 hours | 48 hours
  Electromyography (EMG) is used to measure muscular electrical activity at rest to determine the basal tone. Peak voltage and root mean square (RMS) voltage will be informed.
Surface electromyography at rest - Day 7 | Day 7
  Electromyography (EMG) is used to measure muscular electrical activity at rest to determine the basal tone. Peak voltage and root mean square (RMS) voltage will be informed.
Surface electromyography at maximum voluntary contraction - Baseline | Baseline
  Electromyography (EMG) is used to measure muscular electrical activity at maximum voluntary contraction to determine the recruitment. Peak voltage and RMS voltage will be informed.
Surface electromyography at maximum voluntary contraction - 10 minutes | 10 minutes
  Electromyography (EMG) is used to measure muscular electrical activity at maximum voluntary contraction to determine the recruitment. Peak voltage and RMS voltage will be informed.
Surface electromyography at maximum voluntary contraction - 24 hours | 24 hours
  Electromyography (EMG) is used to measure muscular electrical activity at maximum voluntary contraction to determine the recruitment. Peak voltage and RMS voltage will be informed.
Surface electromyography at maximum voluntary contraction - 48 hours | 48 hours
  Electromyography (EMG) is used to measure muscular electrical activity at maximum voluntary contraction to determine the recruitment. Peak voltage and RMS voltage will be informed.
Surface electromyography at maximum voluntary contraction - Day 7 | Day 7
  Electromyography (EMG) is used to measure muscular electrical activity at maximum voluntary contraction to determine the recruitment. Peak voltage and RMS voltage will be informed.

SECONDARY OUTCOMES:
Visual Analogue Scale of the procedure | Immediately after the intervention
  To determine how unpleasant the procedure is, the visual analog scale (VAS) will be used.
  Expresed in centimeters.
  Minimum value: 0 Maximum value: 10 A higher score implicates a worse outcome.
Post-needling soreness | Four times per day (in the morning, before lunch, in the afternoon, and in the evening) during the seven days following intervention.
  To determine how unpleasant the post-needling soreness is, a pain diary with the visual analog scale (VAS) will be used. The patient will register the pain intensity in the needle area.
  Expresed in centimeters.
  Minimum value: 0 Maximum value: 10 A higher score implicates a worse outcome.
Dose | Immediately after the intervention
  To determine the amount of electric charge applied, the millicoulombs (mC) informed in the MEP device will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Maimónides, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] Girasol CE, Duran NE, D'Almeida SM, Ronzio OA. Toward an algorithm of percutaneous microelectrolysis: a randomized clinical trial on invasive techniques. Sao Paulo Med J. 2025 Aug 11;143(5):e2024164. doi: 10.1590/1516-3180.2024.0164.R1.07032025. eCollection 2025. PMID 40802423